CLINICAL TRIAL: NCT03856658
Title: A Phase II Trial of Hepatic Artery Infusional Floxuridine With Systemic Chemotherapy in the Treatment of Pancreatic Cancer Liver Metastases
Brief Title: Hepatic Artery Infusional Floxuridine to Treat Pancreatic Cancer Liver Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Gerald P. Wright, Surgical Oncology and Hepatopancreaticobiliary Surgeon, Corewell Health West
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-349
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Adenocarcinoma; Liver Metastases
Keywords: pancreatic cancer, pancreatic ductal carcinoma, liver metastases, HAI, hepatic artery infusion pump, FUDR, Floxuridine
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal | interventions — Floxuridine

STUDY DESIGN:
Intervention Model Description: Single arm study without blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Floxuridine (FUDR) via HAI pump (Experimental): Once enrolled, patients will undergo surgical placement of the HAI pump. This can be accomplished using minimally invasive or open techniques with an anticipated hospital stay of approximately 3-5 days. Prior to discharge from the hospital or at the first postoperative visit the pump is filled with FUDR according to the following equation: 0.12 mg/kg/d (using ideal body weight). This fill initiates day 1 of a 4-week cycle. The chemotherapy is infused by the pump continuously over 14 days. On day 15 (+/-4 days), the remaining chemotherapy is removed from the pump which is refilled with heparinized saline (30,000 units). This remains for an additional 2 weeks until the pump is refilled with FUDR at the start of the next cycle. Treatment is continued for a maximum of 6 cycles or as limited by toxicity. This regimen has been utilized with an acceptable safety profile in the setting of colorectal liver metastases.
  Interventions: Drug: Floxuridine (FUDR); Device: Hepatic Artery Infusion Pump; Drug: Heparinized Saline

INTERVENTIONS:
Drug: Floxuridine (FUDR) — Together the FUDR and the HAI pump are experimental because they are being used to treat hepatic liver metastases of Pancreatic adenocarcinoma. They have not yet been FDA approved for this indication, although they are both approved for other indications. The intervention is surgical placement of an HAI pump with subsequent delivery of FUDR via the pump in 28-day cycles. FUDR will be delivered via the HAI pump for 6 months, in 28 day cycles: 2 weeks of therapy, followed by 2 weeks of heparinized saline.
  Other Names: FUDR
Device: Hepatic Artery Infusion Pump — Together the FUDR and the HAI pump are experimental because they are being used to treat hepatic liver metastases of Pancreatic adenocarcinoma. They have not yet been FDA approved for this indication, although they are both approved for other indications. The intervention is surgical placement of an HAI pump with subsequent delivery of FUDR via the pump in 28-day cycles. The primary tumor will be resected or ablated with irreversible electroporation at the time of HAI pump placement. FUDR will be delivered via the HAI pump for 6 months, in 28 day cycles: 2 weeks of therapy, followed by 2 weeks of heparinized saline.
  Other Names: HAI pump; Medtronic pump
Drug: Heparinized Saline — Together the FUDR and the HAI pump are experimental because they are being used to treat hepatic liver metastases of Pancreatic adenocarcinoma. They have not yet been FDA approved for this indication, although they are both approved for other indications. FUDR will be delivered via the HAI pump for 6 months, in 28 day cycles: 2 weeks of therapy, followed by 2 weeks of heparinized saline.

SUMMARY:
This is a single arm, phase II study without blinding. The purpose is to determine the impact of hepatic artery infusion Floxuridine (FUDR) on liver metastases from pancreatic adenocarcinoma. Patients at Spectrum Health will receive standard of care chemotherapy. They will also receive chemotherapy via surgically placed hepatic artery infusion (HAI) pump.

DETAILED DESCRIPTION:
This study hypothesizes that the combination of Floxuridine (FUDR), a type of chemotherapy, delivered via a hepatic artery infusion (HAI) pump, with standard of care systemic chemotherapy will lead to improved survival in the treatment of pancreatic cancer liver metastases. Patients will receive 6 cycles of FUDR and will be followed for two years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proved pancreatic adenocarcinoma with synchronous liver metastases
* Elevated Cancer Antigen 19-9 (CA19-9) at diagnosis (>37 U/mL)
* Ages 18-75 years
* Karnofsky performance status ≥70
* Ability to undergo general anesthesia and HAI pump placement procedure
* CT or MRI scan imaging of the abdomen demonstrating accessibility of the gastroduodenal artery within 2 months of enrollment
* Received a minimum of 2 months of systemic chemotherapy with stable tumor markers and imaging.

Exclusion Criteria:

* Primary tumor resected
* Model for End Stage Liver Disease (MELD) score >20, using the variables of: Bilirubin, serum Sodium, International Normalized Ratio (INR), serum Creatinine, and Dialysis twice in the past week.
* Greater than 60% liver parenchymal involvement by tumor
* Evidence of peritoneal metastases
* Current alcohol abuse
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hepatic progression-free survival | 1 year
  The length of time from the start of trial therapy to the time when target liver lesions show progression or new lesions appear. (Determined by RECIST criteria: ≥20% growth in target lesions and/or appearance of new lesions).

SECONDARY OUTCOMES:
Overall survival | 2 years
  The length of time from diagnosis to death, measured as the proportion of patients surviving at specific time points (6, 12 and 18 months from diagnosis).
Progression-free survival at any site | 2 years
  The length of time from diagnosis to disease progression at any anatomical site (as determined by RECIST criteria) or death.
Rate of tumor response in the liver | 2 years
  Determined by RECIST criteria on imaging studies done every 3 months
EORTC Quality of Life Questionnaire | 2 years
  As measured by the EORTC Quality of Life Questionnaire Core 30 instrument

CONTACTS AND LOCATIONS:
Overall Officials: G. Paul Wright, MD, Principal Investigator — Corewell Health
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No